CLINICAL TRIAL: NCT06548542
Title: A Phase 2a Multicenter, Randomized, Platform Study of Targeted Therapies for the Treatment of Adult Subjects With Moderate to Severe Crohn's Disease
Brief Title: Study of Targeted Therapies for the Treatment of Adult Participants With Moderate to Severe Crohn's Disease
Acronym: Target CD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-885; 2024-513009-30 (Other: EU CT)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Risankizumab; Trosunilimab; Lutikizumab; ABBV-8736
MeSH Terms: conditions — Crohn Disease | interventions — risankizumab; lutikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Monotherapy: Risankizumab (Experimental): Participants will receive Risankizumab Dose A as IV infusion and Risankizumab Dose B as SC injection.
  Interventions: Drug: Risankizumab
- Combination Therapy: Risankizumab and Trosunilimab (Experimental): Participants will receive Risankizumab Dose A as IV infusion and Risankizumab Dose C as SC injection; and trosunilimab Dose A as IV infusion and trosunilimab Dose B as SC injection.
  Interventions: Drug: Risankizumab; Drug: Trosunilimab
- Monotherapy: Trosunilimab (Experimental): Participants will receive trosunilimab Dose A as IV infusion and trosunilimab Dose B as SC injection.
  Interventions: Drug: Trosunilimab
- Combination Therapy: Risankizumab and Lutikizumab (Experimental): Participants will receive Risankizumab Dose A as IV infusion and Risankizumab Dose C as SC injection; and Lutikizumab Dose A, Dose B and Dose C as SC injection.
  Interventions: Drug: Risankizumab; Drug: Lutikizumab
- Monotherapy: Lutikizumab (Experimental): Participants will receive Lutikizumab Dose A, Dose B and Dose C as SC injection.
  Interventions: Drug: Lutikizumab
- Monotherapy: ABBV-8736 - OUS Only (Experimental): Participants will receive ABBV-8736 as IV infusion.
  Interventions: Drug: ABBV-8736
- Long-Term Extension: Risankizumab Monotherapy (Experimental): Participants will receive Risankizumab Dose A as IV infusion and/or Risankizumab Dose B as SC injection for up to 72 weeks.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous Injection
  Arms: Combination Therapy: Risankizumab and Lutikizumab; Combination Therapy: Risankizumab and Trosunilimab; Long-Term Extension: Risankizumab Monotherapy; Monotherapy: Risankizumab
Drug: Lutikizumab — Subcutaneous Injection
  Arms: Combination Therapy: Risankizumab and Lutikizumab; Monotherapy: Lutikizumab
Drug: Trosunilimab — Intravenous Infusion
  Arms: Combination Therapy: Risankizumab and Trosunilimab; Monotherapy: Trosunilimab
Drug: Risankizumab — Intravenous Infusion
  Arms: Combination Therapy: Risankizumab and Lutikizumab; Combination Therapy: Risankizumab and Trosunilimab; Long-Term Extension: Risankizumab Monotherapy; Monotherapy: Risankizumab
Drug: Trosunilimab — Subcutaneous Injection
  Arms: Combination Therapy: Risankizumab and Trosunilimab; Monotherapy: Trosunilimab
Drug: ABBV-8736 — Intravenous Infusion
  Arms: Monotherapy: ABBV-8736 - OUS Only

SUMMARY:
Crohn's disease (CD) is a long-lasting disease that causes severe inflammation (redness, swelling), in the digestive tract, most frequently affecting the bowels. It can cause many different symptoms including belly pain, diarrhea, tiredness, and weight loss. Treatments are available but do not work the same for all patients or may stop working over time. This study will evaluate the effectiveness and adverse events of targeted therapies (TaTs) for adult participants with moderate to severe CD.

The medicines assessed in this study are risankizumab, trosunilimab, lutikizumab, and ABBV-8736. When participants join the study, they will be randomized into available study treatment groups. Adult participants with CD will be enrolled. Around 540 participants will be enrolled in the study at approximately 300 sites worldwide.

Risankizumab and trosunilimab are given as an injection under the skin or as an infusion into the vein. Lutikizumab is given as an injection under the skin. ABBV-8736 is given as an infusion into the vein.

There may be higher treatment burden for participants in this trial compared to their standard of care treatment without participating in this study. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, endoscopies, checking for side effects and completing questionnaires and a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Participants' body weight must be >= 40 kg at Baseline.
* Confirmed diagnosis of CD for at least 3 months prior to Baseline. Documentation of biopsy results consistent with the diagnosis of CD as assessed by the Investigator must be available.
* CDAI >= 220 at Baseline.
* Endoscopic evidence of mucosal inflammation as documented by an SES-CD of >= 6 for ileocolonic or colonic disease or SES-CD of >= 4 for isolated ileal disease. All eligible scores exclude the presence of narrowing component and are determined by a reader.
* Participants must demonstrate intolerance or inadequate response to conventional therapies (OUS) and/or TaTs. TaTs include biologics and/or targeted small molecules.

Exclusion Criteria:

* Participant who demonstrated intolerance to p19 inhibitors, including risankizumab.
* Participant who received any investigational TaT (or TaT that becomes approved during the conduct of the study) within 30 days or 5 half-lives prior to Baseline, whichever is longer. Note: If there is documentation of an undetectable (or below the lower limit of quantification/quantitation) drug level measured by a commercially available assay for any of the approved biologics above, there is no minimum washout prior to Baseline.
* Participant who have any of the following: Current diagnosis of UC or indeterminate colitis. Currently known complications of CD such as: Current ostomy or ileoanal pouch; Current short gut or short bowel syndrome; Surgical bowel resection within the past 3 months prior to Baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Endoscopic Remission | Week 12
  The Simple Endoscopic Score for Crohn's Disease (SES-CD) assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic Remission is defined as SES-CD ≤ 4 and no sub score greater than 1 in any individual variable, as scored by a central reader.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve Endoscopic Response | Week 12
  The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic Response is defined as a decrease in SES-CD ≥ 50% from Baseline, as scored by central reader.
Percentage of Participants With Clinical Remission Per Stool Frequency/Abdominal Pain Score (SF/APS) | Week 12
  SF/APS clinical remission is defined as the average daily SF ≤ 2.8 and not worse than Baseline AND average daily AP score ≤ 1 and not worse than Baseline.
Percentage of Participants With Clinical Remission Per Crohn's Disease Activity Index (CDAI) | Week 12
  The CDAI consists of 8 components; 7 are based on participant diary entries, participant interviews, physical examinations, measurement of body weight and height and 1 is based on laboratory analysis. CDAI clinical remission of Crohn's disease is defined as CDAI < 150

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (254):
- United States (64):
  - Digestive Health Specialists /ID# 266216, Dothan, Alabama
  - East View Medical Research /ID# 270377, Mobile, Alabama
  - Southern California Res. Ctr /ID# 265549, Coronado, California
  - UC San Diego Health System /ID# 265565, La Jolla, California
  - uc davis medical center - patient support services building /ID# 265554, Sacramento, California
  - Clinical Applications Laboratories - San Diego - 3rd Avenue /ID# 267391, San Diego, California
  - Peak Gastroenterology Associates - Colorado Springs - North Cascade Avenue /ID# 265557, Colorado Springs, Colorado
  - Danbury Hospital, Western Connecticut Health Network /ID# 265556, Danbury, Connecticut
  - Yale University School of Medicine /ID# 266786, New Haven, Connecticut
  - Novum Research /ID# 278128, Clermont, Florida
  - University of Florida College of Medicine /ID# 266930, Gainesville, Florida
  - Nature Coast Clinical Research - Inverness /ID# 265874, Inverness, Florida
  - Atlantic Medical Research /ID# 266207, Margate, Florida
  - A Plus Research /ID# 265878, Miami, Florida
  - Sanchez Clinical Research /ID# 265887, Miami, Florida
  - Advanced Research Institute, Inc /ID# 265548, New Port Richey, Florida
  - Hillcrest Medical Research, LLC /ID# 267237, Orange City, Florida
  - Endoscopic Research, Inc. /ID# 267211, Orlando, Florida
  - Gcp Clinical Research /ID# 278126, Tampa, Florida
  - AdventHealth Medical Group - Tampa - Bruce B Downs Boulevard /ID# 265538, Tampa, Florida
  - Florida Medical Clinic - Zephyrhills /ID# 267392, Zephyrhills, Florida
  - Gastroenterology Associates of Central Georgia /ID# 265547, Macon, Georgia
  - Treasure Valley Medical Research /ID# 267114, Boise, Idaho
  - University of Chicago Medical Center /ID# 267400, Chicago, Illinois
  - OSF St. Francis Medical Center /ID# 266973, Peoria, Illinois
  - Springfield Clinic Main Campus /ID# 267434, Springfield, Illinois
  - Indiana University Health University Hospital /ID# 278129, Indianapolis, Indiana
  - University of Kentucky Chandler Medical Center /ID# 265564, Lexington, Kentucky
  - Metropolitan Gastroenterology Group - Chevy Chase /ID# 265877, Chevy Chase, Maryland
  - Lucida Clinical Trials /ID# 266548, New Bedford, Massachusetts
  - Henry Ford Medical Center - Columbus /ID# 266503, Novi, Michigan
  - Mayo Clinic-Rochester /ID# 265550, Rochester, Minnesota
  - GI Associates Research, LLC /ID# 267433, Columbia, Missouri
  - BVL Clinical Research /ID# 265870, Liberty, Missouri
  - Washington University School of Medicine - St. Louis /ID# 266938, St Louis, Missouri
  - Vector Clinical Trials /ID# 265561, Las Vegas, Nevada
  - NYU Langone Long Island Clinical Research Association /ID# 265566, Great Neck, New York
  - Icahn School of Medicine at Mount Sinai /ID# 266857, New York, New York
  - Northwell Health-Lenox Hill Hospital /ID# 265527, New York, New York
  - Care Access - Yonkers /ID# 266781, Yonkers, New York
  - Digestive Health Partners - Biltmore Office /ID# 265539, Asheville, North Carolina
  - Velocity Clinical Research - Durham /ID# 267712, Durham, North Carolina
  - University of Cincinnati /ID# 265589, Cincinnati, Ohio
  - The Ohio State University /ID# 265577, Columbus, Ohio
  - Digestive Disease Specialists - Oklahoma /ID# 265901, Oklahoma City, Oklahoma
  - Penn State Health Milton South Hershey Medical Center /ID# 267126, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 265904, Philadelphia, Pennsylvania
  - Gastroenterology Associates of Orangeburg /ID# 267548, Orangeburg, South Carolina
  - GI associates of Northeast Tennessee /ID# 265567, Johnson City, Tennessee
  - Gi Alliance - Cedar Park /ID# 268153, Cedar Park, Texas
  - Proactive Clinical Research /ID# 267305, El Paso, Texas
  - Digestive Health Associates of Texas (DHAT) Research Institute - Garland /ID# 266935, Garland, Texas
  - Houston Methodist Hospital /ID# 265533, Houston, Texas
  - Caprock Gastro Research - Lubbock - 80th Street /ID# 265541, Lubbock, Texas
  - GI Alliance: Mansfield /ID# 266947, Mansfield, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 265899, San Antonio, Texas
  - Sun Research Institute /ID# 266723, San Antonio, Texas
  - Southern Star Research Institute /ID# 278124, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake /ID# 265576, Southlake, Texas
  - Tyler Research Institute, LLC /ID# 265545, Tyler, Texas
  - Care Access - Ogden /ID# 266428, Ogden, Utah
  - Care Access - Salt Lake City /ID# 266785, Salt Lake City, Utah
  - Virginia Mason Hospital & Medical Center /ID# 265574, Seattle, Washington
  - Washington Gastroenterology - Tacoma /ID# 267302, Tacoma, Washington
- Austria (6):
  - Medizinische Universitaet Graz /ID# 275453, Graz, Styria
  - Medizinische Universitaet Innsbruck /ID# 265930, Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 265929, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH /ID# 266035, Wels, Upper Austria
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 265928, Salzburg
  - Medizinische Universitaet Wien /ID# 265926, Vienna
- Belgium (10):
  - Imelda Ziekenhuis /ID# 265995, Bonheiden, Antwerpen
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 265993, Anderlecht, Brussels Capital
  - CHU Saint-Pierre /ID# 266431, Brussels, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 265521, Brussels, Brussels Capital
  - Groupe Sante CHC - Clinique du MontLegia /ID# 265522, Liège, Liege
  - Universite Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant /ID# 265517, Yvoir, Namur
  - UZ Leuven /ID# 265519, Leuven, Vlaams-Brabant
  - AZ Groeninge /ID# 265544, Kortrijk, West-Vlaanderen
  - AZ Oostende /ID# 275534, Ostend, West-Vlaanderen
  - CHU de Liege /ID# 265542, Liège
- Bulgaria (8):
  - Hospital Tsaritsa Yoanna /ID# 266235, Sofiya, Sofia
  - Medical Center - Doverie /ID# 267050, Sofiya, Sofia
  - ACIBADEM City Clinic Diagnostic-Consultative Center /ID# 266239, Sofiya, Sofia
  - Umbal Kaspela /ID# 266234, Plovdiv
  - MHAT Knyaginya Klementina /ID# 266238, Sofia
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 267437, Sofia
  - Military Medical Academy Multiprofile Hospital /ID# 267051, Sofia
  - UMHAT Multiprofile Hospital for Active Treatment Sveta Marina /ID# 266237, Varna
- Canada (8):
  - University of Calgary /ID# 265524, Calgary, Alberta
  - Gastroenterology and Internal Medicine Research Institute /ID# 265610, Edmonton, Alberta
  - University of Alberta Hospital /ID# 265614, Edmonton, Alberta
  - Medicor Research /ID# 267405, Greater Sudbury, Ontario
  - London Health Sciences Centre - University Hospital /ID# 267298, London, Ontario
  - Toronto Digestive Disease Associates /ID# 267358, Vaughan, Ontario
  - Clinique IMD /ID# 272057, Montreal, Quebec
  - Diex Recherche Quebec Inc. /ID# 265611, Québec
- Croatia (5):
  - Klinicki Bolnicki Centar Zagreb /ID# 265502, Grad Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 265509, Zagreb, City of Zagreb
  - Poliklinika Borzan d.o.o. /ID# 265503, Osijek, County of Osijek-Baranja
  - Specialty Hospital Medico /ID# 265504, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 265511, Split, Split-Dalmatia County
- Czechia (3):
  - Hepato-Gastroenterologie HK /ID# 265387, Hradec Králové, Hradec Kralove
  - Iscare Klinické Centrum /ID# 265407, Prague, Praha 9
  - SurGal Clinic /ID# 265388, Brno, South Moravian
- Denmark (2):
  - Aarhus Universitetshospital - Skejby /ID# 269064, Aarhus, Central Jutland
  - Odense University Hospital /ID# 267778, Odense, Region Syddanmark
- Estonia (3):
  - Medicum /ID# 268304, Tallinn, Harju
  - East Tallinn Central Hospital /ID# 267658, Tallinn
  - Tartu University Hospital /ID# 267656, Tartu
- Finland (2):
  - Tampere University Hospital /ID# 267721, Tampere, Pirkanmaa
  - Turku University Hospital /ID# 267723, Turku, Southwest Finland
- France (10):
  - Chu de Nice-Hopital Larchet Ii /Id# 267478, Nice, Alpes-Maritimes
  - CHU de Toulouse - Hôpital Rangueil /ID# 267479, Toulouse, Haute-Garonne
  - CHU de Montpellier - Hopital Saint Eloi /ID# 265718, Montpellier, Herault
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou /ID# 266848, Rennes, Ille-et-Vilaine
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois /ID# 265703, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Hospitalier Universitaire de Bordeaux /ID# 265721, Pessac, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 265340, St-Priest-en-Jarez, Pays de la Loire Region
  - Hospices Civils de Lyon - Centre Hospitalier Lyon-Sud /ID# 266851, Pierre-Bénite, Rhone
  - Clinique Jules Verne /ID# 267480, Nantes
  - Hopital Saint Antoine /ID# 265725, Paris
- Germany (20):
  - Universitaetsklinikum Freiburg /ID# 265755, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsmedizin Mannheim /ID# 266961, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 266962, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 265927, Erlangen, Bavaria
  - Klinikum der Universitaet Muenchen Grosshadern /ID# 269165, Munich, Bavaria
  - Markus Krankenhaus /ID# 265938, Frankfurt am Main, Hesse
  - Universitaetsklinikum Frankfurt /ID# 266827, Frankfurt am Main, Hesse
  - Klinikum Lueneburg /ID# 266886, Lüneburg, Lower Saxony
  - Universitaetsmedizin Essen /ID# 275535, Essen, North Rhine-Westphalia
  - St. Marien- und St. Annastiftskrankenhaus /ID# 265912, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Universitaetsklinikum des Saarlandes /ID# 265753, Homburg, Saarland
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 265931, Dresden, Saxony
  - Eugastro /ID# 266826, Leipzig, Saxony
  - Studiengesellschaft BSF Unternehmergesellschaft /ID# 265751, Halle, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel /ID# 265738, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck /ID# 267254, Lübeck, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 265752, Berlin
  - DRK Kliniken Berlin - Westend /ID# 265925, Berlin
  - Krankenhaus Waldfriede /ID# 266676, Berlin
  - Universitaetsklinikum Regensburg /ID# 275556, Regensburg
- Hungary (6):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 267389, Debrecen, Hajdú-Bihar
  - Clinfan /ID# 267385, Szekszárd, Tolna County
  - Synexus Hungary Clinical Research Centre - Budapest /ID# 267384, Budapest
  - Semmelweis Egyetem /ID# 267064, Budapest
  - Semmelweis Egyetem /ID# 267068, Budapest
  - Szegedi Tudomanyegyetem /ID# 267386, Szeged
- Ireland (7):
  - Letterkenny General Hospital /ID# 276677, Letterkenny, Donegal
  - Portiuncula University Hospital /ID# 267771, Ballinasloe, Galway
  - Our Lady of Lourdes Hospital - Drogheda /ID# 267768, Drogheda, Louth
  - Midland Regional Hospital Mullingar /ID# 267769, Mullingar, Westmeath
  - St. Vincent's University Hospital /ID# 267766, Dublin
  - Beaumont Hospital /ID# 267770, Dublin
  - Connolly Hospital /ID# 268021, Dublin
- Israel (4):
  - Edith Wolfson Medical Center /ID# 267640, Holon, Central District
  - Soroka Medical Center /ID# 267235, Beersheba, Southern District
  - Tel Aviv Sourasky Medical Center /ID# 267307, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus- Haifa /ID# 267641, Haifa
- Italy (11):
  - Azienda Ospedaliero Universitaria di Cagliari - P.O. Duilio Casula /ID# 267287, Monserrato, Cagliari
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 267143, San Giovanni Rotondo, Foggia
  - IRCCS Istituto Clinico Humanitas /ID# 265946, Rozzano, Lombardy
  - IRCCS Ospedale San Raffaele /ID# 265951, Milan, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 265935, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 265940, Rome, Roma
  - A.O. Ordine Mauriziano di Torino /ID# 267144, Turin, Torino
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 265942, Negrar, Verona
  - Azienda Ospedaliero-Universitaria Renato Dulbecco /ID# 267722, Catanzaro
  - Azienda Ospedaliera Universitaria Gaetano Martino /ID# 267145, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 265949, Milan
- Latvia (3):
  - Liepaja Regional Hospital /ID# 267703, Liepāja
  - Pauls Stradins Clinical University Hospital /ID# 267705, Riga
  - Digestive Diseases Center GASTRO /ID# 267707, Riga
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 267695, Kaunas
  - Panevezys Republican Hospital /ID# 267709, Panevezys
  - Vilnius University Hospital Santaros Klinikos /ID# 267711, Vilnius
- Netherlands (4):
  - Elisabeth TweeSteden Ziekenhuis /ID# 265729, Tilburg, North Brabant
  - Amsterdam UMC, locatie AMC /ID# 268321, Amsterdam, North Holland
  - Universitair Medisch Centrum Groningen /ID# 265736, Groningen
  - Universitair Medisch Centrum Utrecht /ID# 265731, Utrecht
- Norway (3):
  - Akershus University Hospital /ID# 267642, Lørenskog, Akershus
  - Helse More- og Romsdal HF, Alesund sjukehus /ID# 267632, Ålesund, Møre og Romsdal
  - Oslo Universitetssykehus Ulleval /ID# 267630, Oslo
- Poland (8):
  - NZOZ Centrum Medyczne KERmed /ID# 266766, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Gastromed Sp. z o.o /ID# 266765, Torun, Kuyavian-Pomeranian Voivodeship
  - Malopolskie Centrum Kliniczne /ID# 265943, Krakow, Lesser Poland Voivodeship
  - Medical Network Sp.z.o.o. WIP Warsaw IBD Point Profesor Kierkus /ID# 266764, Warsaw, Masovian Voivodeship
  - Bodyclinic Sp. z o.o. sp.k. /ID# 265945, Warsaw, Masovian Voivodeship
  - Endoskopia Sp. z.o.o. /ID# 265934, Sopot, Pomeranian Voivodeship
  - H-T Centrum Medyczne Endoterapia /ID# 265937, Tychy, Silesian Voivodeship
  - Polimedica PTG Kielce /ID# 267066, Kielce, Świętokrzyskie Voivodeship
- Portugal (6):
  - Unidade Local de Saude do Alto Ave, EPE /ID# 265892, Guimarães, Braga District
  - 2CA-Braga, Hospital de Braga /ID# 265894, Braga
  - Unidade Local de Saude de Coimbra, EPE /ID# 267240, Coimbra
  - Unidade Local de Saude de Lisboa Ocidental, EPE /ID# 267242, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE /ID# 266113, Lisbon
  - Unidade Local de Saude do Alto Minho, EPE - Hospital de Santa Luzia /ID# 265885, Viana do Castelo
- Romania (4):
  - Memorial Healthcare International S.R.L. /Id# 267328, Bucharest, București
  - Spitalul Clinic Colentina /ID# 267208, Bucharest, București
  - Clinica Gastro Med SRL /ID# 267204, Cluj-Napoca, Cluj
  - OncoHelp Association /ID# 267203, Timișoara, Timiș County
- Serbia (7):
  - Clinical Hospital Center Zvezdara /ID# 265605, Belgrade, Beograd
  - Military Medical Academy /ID# 267452, Belgrade, Beograd
  - University Clinical Hospital Center "Dr. Dragisa Misovic - Dedinje" /ID# 265607, Belgrade, Beograd
  - Clinical Hospital Center - Bežanijska Kosa /ID# 265604, Belgrade, Beograd
  - Leskovac General Hospital /ID# 265606, Leskovac, Jablanicki Okrug
  - General Hospital Djordje Joanovic /ID# 266040, Zrenjanin, Vojvodina
  - University Clinical Center Vojvodina /ID# 265603, Novi Sad
- Singapore (3):
  - Mount Elizabeth Hospital /ID# 268354, Singapore, Central Singapore
  - Gleneagles Hospital /ID# 268385, Singapore, Central Singapore
  - National University Hospital /ID# 268128, Singapore
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 266064, Banská Bystrica, Banská Bystrica Region
  - KM Management, spol. s.r.o. /ID# 266070, Nitra, Nitra Region
  - Gastro I., s.r.o. /ID# 267159, Prešov, Presov
  - ENDOMED s.r.o /ID# 266068, Košice
- Slovenia (2):
  - General Hospital Celje /ID# 267699, Celje
  - University Medical Centre Ljubljana /ID# 267697, Ljubljana
- South Korea (6):
  - Inje University Haeundae Paik Hospital /ID# 266380, Busan, Busan Gwang Yeogsi
  - Dong-A University Medical Center /ID# 266709, Busan, Busan Gwang Yeogsi
  - The Catholic University of Korea, Daejeon St. Mary's Hospital /ID# 265488, Daejeon, Daejeon Gwang Yeogsi
  - Chungang University Hospital /ID# 266427, Dongjak-gu, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 265489, Seoul, Seoul Teugbyeolsi
  - Kyungpook National University Chilgok Hospital /ID# 265487, Daegu
- Spain (8):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 266902, Santiago de Compostela, A Coruna
  - Hospital Universitario Virgen Macarena /ID# 266648, Seville, Sevilla
  - Hospital Universitario Virgen del Rocio /ID# 266727, Seville, Sevilla
  - Hospital Clinic de Barcelona /ID# 265415, Barcelona
  - Hospital Universitario 12 de Octubre /ID# 265444, Madrid
  - Hospital Universitario La Paz /ID# 265412, Madrid
  - Hospital Alvaro Cunqueiro /ID# 266647, Pontevedra
  - Hospital Universitari i Politècnic La Fe /ID# 265478, Valencia
- Switzerland (3):
  - University Hospital Zurich /ID# 275755, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 265733, Bern
  - Intesto /ID# 265728, Bern
- Taiwan (4):
  - China Medical University Hospital /ID# 265924, Taichung
  - National Taiwan University Hospital /ID# 265921, Taipei
  - Taipei Veterans General Hospital /ID# 276064, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 265922, Taoyuan
- Turkey (Türkiye) (5):
  - Kocaeli University Research and Application Hospital /ID# 267772, Dilovası, Kocaeli
  - Hacettepe Universitesi Tip Fakultesi /ID# 266394, Ankara
  - Bezmialem Vakif Üniversitesi /ID# 266399, Istanbul
  - Istanbul University Istanbul Medical Faculty /ID# 266299, Istanbul
  - Karadeniz Teknik Universitesi Tip Fakultesi /ID# 266303, Trabzon
- United Kingdom (12):
  - Western General Hospital - NHS Lothian /ID# 266333, Edinburgh, Edinburgh, City of
  - Gartnavel General Hospital /ID# 266407, Glasgow, Glasgow City
  - Barts Health NHS Trust /ID# 266410, London, Greater London
  - Royal Free Hospital /ID# 268065, London, Greater London
  - Guy's Hospital /ID# 266336, London, Greater London
  - St George University Hospitals NHS Foundation Trust /ID# 266335, London, Greater London
  - The John Radcliffe Hospital /ID# 266334, Oxford, Oxfordshire
  - The Royal Wolverhampton NHS Trust /ID# 268158, Guildford, Surrey
  - University Hospital Coventry & Warwickshire NHS Trust /ID# 267128, Coventry, Warwickshire
  - Velocity Clinical Research - Bristol /ID# 275736, Bristol
  - University Hospital of Wales /ID# 275702, Cardiff
  - Royal Victoria Infirmary /ID# 268064, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-885